CLINICAL TRIAL: NCT06505408
Title: Evaluating the Impact of a Multivitamin Supplement to Support Biomarkers Associated With Conception and Pregnancy in Healthy Women
Brief Title: Impact of a MVM to Support Biomarkers Associated With Conception and Pregnancy in Healthy Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perelel Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AFRCO-182
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Healthy Adult Women of Child Bearing Age
Keywords: Multivitamin; Healthy women
MeSH Terms: interventions — Geritol

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, placebo-controlled, parallel study in healthy women.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Multivitamin (Experimental)
  Interventions: Dietary Supplement: Multivitamin

INTERVENTIONS:
Dietary Supplement: Multivitamin — 4 capsules of Perelel Health Conception Support Multivitamin Pack (consisting of vitamins, minerals, and omega ingredients) consumed daily for 12 weeks
  Other Names: MVM
  Arms: Multivitamin
Dietary Supplement: Placebo — 4 placebo capsules consumed daily for 12 weeks
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the effects multivitamin (MVM) on blood biomarkers that are associated with healthy pregnancy and conception in adult women. The main question it aims to answer is:

Is there a significant change in blood biomarkers from baseline (week 0) to end of intervention (week 12) in healthy women consuming multivitamin compared to participants consuming the placebo product?

Participants will:

Take drug MVM or a placebo every day for 12 weeks Visit the clinic at baseline and 12 weeks for serum blood draws and measurements Complete a series of surveys at baseline and 12 weeks

DETAILED DESCRIPTION:
A 12 week double-blind, placebo-controlled, clinical trial assessing the daily administration of a multivitamin (MVM) or placebo on blood biomarkers associated with healthy pregnancy and conception in healthy adult women. Participants will consume study product or placebo for 12 weeks. Measurements will be taken at baseline and at the end of 12 weeks.

Primary Objective: To evaluate in healthy women, the effect of 12-week long daily administration of a multivitamin (MVM) on blood biomarkers associated with healthy pregnancy (Folate).

Secondary Objective: To evaluate in healthy women, the effect of 12-week long daily administration of multivitamin (MVM) on blood biomarkers associated with healthy pregnancy

* Vitamin B12
* Iron
* Omega-3
* Choline
* CoQ10

ELIGIBILITY:
Inclusion Criteria:

* Be able to give written informed consent.
* Be between 21- 40 years of age (inclusive).
* Regular menstrual cycles in the past 6 months.
* Willing to consume the study product daily for the duration of the study.

Exclusion Criteria:

* Participants who are pregnant or wish to become pregnant during the study or who are lactating and/or currently breastfeeding.
* Participants currently of biological childbearing potential, but not using a continuous effective method of contraception, as outlined below:

  1. Complete abstinence from intercourse two weeks prior to administration of the Study Product, throughout the clinical study, until the completion of follow-up procedures or for two weeks following discontinuation of the Study Product in cases where Participant discontinues the study prematurely. (Participants utilizing this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding two weeks when they present to the clinic for the final visit).
  2. Has a male sexual partner who is surgically sterilised prior to the Screening Visit and is the only male sexual partner for that Participant.
  3. Sexual partner(s) is/are exclusively female.
  4. Use of acceptable method of contraception, such as a spermicide, mechanical barrier (e.g., male condom, female diaphragm), tubal ligation. The Participant must be using this method for at least one week prior to and one week following the end of the study.
* Has a history of drug and/or alcohol abuse at the time of enrolment.
* Is a smoker.
* Is hypersensitive to any of the contents of the study product, that would preclude intake of the study products.
* Has any significant acute or chronic coexisting health conditions that would prevent them from fulfilling the study requirements, put the Participant at risk or would confound the interpretation of the study results as judged by the investigator on the basis of medical history.

Excluded health conditions include:

a. Diabetes mellitus b. Cardiovascular disease c. Class II/III obesity (defined as BMI ≥35.0 Kg/m2)

* Current or recent (in the past 12 weeks) use of a medication that the investigator believes would interfere with the objectives of the study or pose a safety risk or confound the interpretation of the study results. Prohibited medications include:

  a. Oral contraceptive pills
* Current or recent (in the past 4 weeks) use of prohibited nutritional or non-nutritional supplements, including:

  a. Vitamins/minerals (vitamin D, folate, vitamin B12)
* Current or recent (in the past 8 weeks) use of prohibited nutritional or non-nutritional supplements, including:

  1. Omega supplements
  2. Iron
* Individuals who, in the opinion of the investigator, are considered to be poor
* If the Participant has been in a recent experimental study involving drugs/supplements, these must have been completed not less than 90 days for drugs and 30 days for supplements prior to this study.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 60 (Actual)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline (week 0) to end of intervention (week 12) on Serum Folate | 12 weeks

SECONDARY OUTCOMES:
Change from baseline (week 0) to end of intervention (week 12) on Serum Iron [including Ferritin, Total Iron Binding Capacity (TIBC) and Transferrin] | 12 weeks
Change from baseline (week 0) to end of intervention (week 12) on Serum Vitamin B12 | 12 weeks
Change from baseline (week 0) to end of intervention (week 12) on Ratio Omega 6: Omega 3 (calculated) | 12 weeks
Change from baseline (week 0) to end of intervention (week 12) on RBC Fatty Acid of Omega-3(DHA and EPA) and Omega-6 (CLA and AA) | 12 weeks
Change from baseline (week 0) to end of intervention (week 12) on plasma Choline | 12 weeks
Change from baseline (week 0) to end of intervention (week 12) on plasma CoQ10 | 12 weeks
Change from baseline (week 0) to end of intervention (week 12) on serum C-Reactive Protein (CRP) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dinan, MD, PHD, Principal Investigator — Atlantia Clinical Trials
Locations (1):
- Atlantia Food Clinical Trials, Cork, Munster, Ireland

IPD SHARING:
Plan to Share IPD: No